CLINICAL TRIAL: NCT05534503
Title: Is it Necessary to Drain in Contact With the Prostheses During a Cure of a Ventricle With Retromuscular Prosthesis?
Acronym: Drain-IHR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8704
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Eventration of the Abdominal Wall
Keywords: Eventration of the abdominal wall; Hernia; Drainage; Retromuscular position; Digestive surgery
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Is there an indication for drainage in contact with a prosthesis placed in a retromuscular position, during a cure for abdominal wall ventration in adults? This procedure is very frequent in digestive surgery and can be associated with serious complications, notably prosthesis infection.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Patient operated on at HUS between 01/01/2018 and 12/31/2020
* Patient who has undergone surgical cure of anterior or lateral abdominal wall eventration of any width with placement during the procedure of a prosthetic mesh in a prefascial retromuscular position.
* Patient not objecting to the reuse of their data for scientific research purposes.

Exclusion criteria:

* Patient who has expressed opposition to the reuse of his or her data for scientific research purposes.
* Particular clinical forms of the disease: absence of previous surgical intervention (and thus absence of ventration: umbilical hernia, diastasis)
* Absence of prosthesis during the operation or prosthesis placed in intraperitoneal position

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) operated on at HUS between 01/01/2018 and 12/31/2020
Sampling Method: Non-Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2022-07-31 (Actual); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
infection after drainage in contact with a retromuscular prosthesis | 1 day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Service de chirurgie générale et digestive - CHU de Strasbourg - France, Strasbourg, France